CLINICAL TRIAL: NCT03039985
Title: All-ceramic Crowns in Patients With Sleep Bruxism - a Randomized Clinical Trial
Brief Title: All-ceramic Crowns in Patients With Sleep Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Brigitte Ohlmann, Prof. Dr. med.dent., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCHM2456/4-1
Record Dates: First submitted 2017-01-13; First posted 2017-02-01 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Sleep Bruxism; Monolithic Ceramic Fixed Dental Prosthesis (Single Crowns)
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Bruxism + lithium disilicate crown (Experimental): Participant with sleep bruxism receives a monolithic molar crown manufactured from lithium disilicate.
  Interventions: Device: lithium disilicate crowns (IPSe.max®)
- No bruxism + lithium disilicate crown (Experimental): Participant without sleep bruxism receives a monolithic molar crown manufactured from lithium disilicate.
  Interventions: Device: lithium disilicate crowns (IPSe.max®)
- Bruxism + zirconia crown (Experimental): Participant with sleep bruxism receives a monolithic molar crown manufactured from zirconia.
  Interventions: Device: Zirconia crowns (Prettau®)
- No bruxism + zirconia crown (Experimental): Participant without sleep bruxism receives a monolithic molar crown manufactured from zirconia.
  Interventions: Device: Zirconia crowns (Prettau®)

INTERVENTIONS:
Device: Zirconia crowns (Prettau®) — Monolithic zirconia molar crowns are, after randomization, placed in patients with or without bruxism
  Arms: Bruxism + zirconia crown; No bruxism + zirconia crown
Device: lithium disilicate crowns (IPSe.max®) — lithium disilicate molar crowns are, after randomization, placed in patients with or without bruxism
  Arms: Bruxism + lithium disilicate crown; No bruxism + lithium disilicate crown

SUMMARY:
The aim of the study is to evaluate the complication rate of 2 types of all-ceramic crowns in patients with or without bruxism.

ELIGIBILITY:
Inclusion Criteria:

* need a molar crown
* tooth antagonist (no implant)

Exclusion Criteria:

* no Antagonist pregnancy, bleeding, periodontal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-02; Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Success of all-ceramic crowns as determined by complication rate | up to 5 years
  In this study, a complication is defined as any event happening at the study crown or the supporting tooth that requires a clinical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Ohlmann, Prof. Dr., Principal Investigator — Heidelberg University; Marc Schmitter, Prof. Dr., Principal Investigator — University of Würzburg
Locations (1):
- Department of Prosthodontics, University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Ohlmann B, Rathmann F, Bomicke W, Behnisch R, Rammelsberg P, Schmitter M. Validity of patient self-reports and clinical signs in the assessment of sleep bruxism based on home-recorded electromyographic/electrocardiographic data. J Oral Rehabil. 2022 Jul;49(7):720-728. doi: 10.1111/joor.13327. Epub 2022 Apr 11. PMID 35348247
- [Derived] Ohlmann B, Bomicke W, Behnisch R, Rammelsberg P, Schmitter M. Variability of sleep bruxism-findings from consecutive nights of monitoring. Clin Oral Investig. 2022 Apr;26(4):3459-3466. doi: 10.1007/s00784-021-04314-8. Epub 2021 Dec 3. PMID 34862565
- [Derived] Ohlmann B, Bomicke W, Habibi Y, Rammelsberg P, Schmitter M. Are there associations between sleep bruxism, chronic stress, and sleep quality? J Dent. 2018 Jul;74:101-106. doi: 10.1016/j.jdent.2018.05.007. Epub 2018 May 17. PMID 29777735